CLINICAL TRIAL: NCT02377154
Title: Comparability of Keratometry and Intraocular Lens (IOL) Calculation of VERION Image Guided System With Established Measuring Devices in Ophthalmologically Healthy Individuals
Brief Title: Comparability of Keratometry of VERION Image Guided System With Established Measuring Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Mike P. Holzer, Ophthalmologist, FEBO, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-532/2014
Record Dates: First submitted 2015-02-13; First posted 2015-03-03 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: keratometry; verion; iol; intraocular lens; iolmaster; lenstar; pentacam; IOL calculation; VERION Image Guided System
MeSH Terms: conditions — Intraocular Lymphoma | interventions — Slit Lamp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Opthalmologically healthy individuals (Other): Slit lamp, Autorefractor, IOLMaster 500, Pentacam HR, LenStar LS900, VERION Image Guided System
  Interventions: Device: Slit lamp; Device: Autorefractor; Device: IOLMaster 500; Device: Pentacam HR; Device: LenStar LS900; Device: VERION Image Guided System

INTERVENTIONS:
Device: Slit lamp — Examination of cornea
Device: Autorefractor — Measurement of refraction
Device: IOLMaster 500 — Measurement of axial length and white-to-white distance; Keratometry; IOL calculation
Device: Pentacam HR — Measurement of white-to-white distance; Keratometry
Device: LenStar LS900 — Measurement of axial length and white-to-white distance; Keratometry; IOL calculation
Device: VERION Image Guided System — Measurement of white-to-white distance; Keratometry; IOL calculation with axial length value of IOLMaster 500

SUMMARY:
The purpose of this study is to determine if the keratometric functions of the VERION Image Guided System are comparable to those of established keratometric devices (IOLMaster 500, Pentacam HR, LenStar LS900). Calculated intraocular lenses (IOLs) are compared as a clinical consequence of the biometric measurement for IOLMaster 500, LenStar LS900 and VERION Image Guided System.

In addition the comfort and duration of examination in the different devices is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All interested individuals
* Full legal capacity

Exclusion Criteria:

* Pre-existing or actual ocular disease or pathology, history of ocular surgery
* Contact lens wear 2 weeks before examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of repeatability of keratometry as performed by VERION Image Guided System | 3 immediate repetitions at study visit (study consists of 1 visit only)

SECONDARY OUTCOMES:
Subjective comfort for test persons as evaluated by questionnaire | Immediately after study visit (study consists of 1 visit only)
Duration of measurements of each keratometric device as taken by stopwatch | During measurements from placement of head until completion
Keratometric values as measured by IOLMaster 500, Pentacam HR, LenStar LS900, VERION Image Guided System | At study visit (study consists of 1 visit only)
White-to-White distance as measured by IOLMaster 500, Pentacam HR, LenStar LS900, VERION Image Guided System | At study visit (study consists of 1 visit only)
Intraocular lens calculation as performed by IOLMaster 500, LenStar LS900, VERION Image Guided System | Immediately after measurement

CONTACTS AND LOCATIONS:
Overall Officials: Mike P Holzer, MD, FEBO, Principal Investigator — Department of opthalmology, University of Heidelberg
Locations (1):
- Department of ophthalmology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany